CLINICAL TRIAL: NCT07269015
Title: Evaluation of the Accuracy of Continuous Glucose Monitoring Systems and Educational Needs in Pregnant Women With Diabetes: A Comparison Between Dexcom One Plus and FreeStyle Libre 2 Plus
Brief Title: CGM Accuracy in Pregnancy Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P/25-041
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Pregestational Diabetes; Continuous Glucose Monitoring
Keywords: type 2 diabetes; continuous glucose monitoring; pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: All participants receive both sensors simultaneously
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dual Continuous Glucose Monitoring Use (Experimental): All participants will wear two continuous glucose monitoring sensors simultaneously
  Interventions: Device: Dexcom One Plus; Device: FreeStyle Libre 2 Plus; Procedure: Additional Study Procedures

INTERVENTIONS:
Device: Dexcom One Plus — Worn on the upper arm for 10 days Two replacements during the 30-day study period Used with Dexcom mobile application
Device: FreeStyle Libre 2 Plus — Worn on the opposite arm for 15 days One replacement during the 30-day study period Used as real-time CGM via LibreLink
Procedure: Additional Study Procedures — Capillary glucose monitoring before meals, 1 hour postprandially, and during symptoms of hypoglycemia (Contour Instant) One baseline structured education session for participants without prior CGM experience Routine diabetes education according to national guidelines

SUMMARY:
Pregnancy in women with diabetes remains a high-risk condition, requiring strict glycemic control due to rapid physiological changes that affect insulin sensitivity. Continuous glucose monitoring (CGM) provides detailed glucose trends, but the accuracy of newer, affordable systems such as Dexcom One Plus and FreeStyle Libre 2 Plus has not been evaluated during pregnancy.

This prospective interventional study aims to compare the accuracy of these two CGM systems-both worn simultaneously-using capillary glucose as the reference. The study also evaluates educational needs, skills, attitudes, digital competence, lifestyle habits, and patient-reported outcomes among pregnant women with type 1 diabetes (T1D), type 2 diabetes (T2D), and gestational diabetes (GDM).

DETAILED DESCRIPTION:
Women with diabetes during pregnancy experience increased risks of congenital malformations, neonatal morbidity, hypertensive disorders, and abnormal fetal growth. Continuous glucose monitoring (CGM) improves glycemic outcomes in type 1 diabetes (T1D) in pregnancy, yet evidence remains limited for type 2 diabetes (T2D) and gestational diabetes (GDM). Dexcom One Plus and FreeStyle Libre 2 Plus are recent low-cost systems with CE-mark approval for use in pregnancy, both with reported Mean Absolute Relative Difference (MARD) values around 8%. However, neither system has been specifically validated in pregnant populations.

Physiological changes in pregnancy-including increased total body water and interstitial fluid-may alter CGM accuracy. Prior studies show that earlier FreeStyle Libre versions may overestimate hypoglycemia in pregnant women. Furthermore, women with T2D or GDM typically have little prior exposure to diabetes education or CGM technology, which may contribute to suboptimal glycemic control.

This study evaluates the accuracy and usability of Dexcom One Plus and FreeStyle Libre 2 Plus during pregnancy, while also assessing educational and digital literacy needs to optimize CGM implementation in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with type 1 diabetes, type 2 diabetes, or gestational diabetes, diagnosed before 32 weeks of gestation
* Age ≥18 years
* Willingness to wear two CGM systems simultaneously
* Possession of a smartphone compatible with LibreLink
* Ability to sign informed consent

Exclusion Criteria:

* Comorbidities affecting glucose metabolism
* Inability to use CGM devices or perform capillary glucose testing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Mean Absolute Relative Difference (MARD) | End of 30-day monitoring period; Primary outcome
  Difference between paired continuous glucose monitoring (CGM) readings (Dexcom One Plus vs. FreeStyle Libre 2 Plus) and reference capillary glucose values.
Baseline diabetes knowledge, skills, and attitudes | Baseline (first study visit)
  For the baseline evaluation, a specific questionnaire for the present study was administered, and the Spanish version of the Cambados Questionnaire will also be used. The Cambados Questionnaire is a 5-item questionnaire designed to assess digital competence. The score range is from 0 to 20. Higher scores indicate greater digital competence.

SECONDARY OUTCOMES:
Mean Absolute Difference (MAD) for glucose <70 mg/dL | End of 30-day monitoring period
  |Difference| between paired values.
Agreement rates (15/15%, 20/20%, 40/40%) across glucose ranges | End of 30-day monitoring period
  Categories: <63, 63-140, <70, 70-180, >140, >180 mg/dL.
Dietary habits (Mediterranean diet adherence) | Baseline and End of 30-day monitoring period
  The Mediterranean Diet Adherence Screener (MEDAS) will be used to evaluate adherence to the Mediterranean diet using a 17-item dietary assessment (score range: 0-17). Higher scores indicate greater adherence to the Mediterranean diet.
Physical activity | 7 days before baseline and through study completion, an average of 1 week
  Physical activity will be assessed by steps per day (measured as total steps) and using the reduced version of the Pregnancy Physical Activity Questionnaire (PPAQ). The reported time spent in each activity category will be multiplied by the established categorical intensity value (METs) associated with that question. The total weekly physical activity level (MET-minutes/week or MET-hours/week) will be calculated by summing the MET values for each item, allowing for classification by intensity (sedentary, light, moderate, and vigorous)
Sleep quality | Baseline and through study completion, an average of 1 week
  Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-item, self-rated questionnaire designed to measure sleep quality and disturbance. Sleep component scores will be summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality
Patient-reported outcomes (PROMs) | Through study completion, an average of 1 week
  The Glucose Monitoring System Satisfaction Survey (GMSS) will be used to assess patients' satisfaction with their continuous glucose monitoring (CGM) system. GMSS is a 15-item questionnaire with a score range of 1 to 5. Higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Driesman AS, Konopka JA, Feder O, Aggarwal V, Schwarzkopf R. Management Principles of Massive Acetabular Bone Loss in Revision Total Hip Arthroplasty A Review of the Literature. Bull Hosp Jt Dis (2013). 2023 Mar;81(1):4-10. PMID 36821729
- [Background] Dai J, Liu D, Yin X, Wen X, Cai G, Zheng L. Anisotropic Elastomer Ionomer Composite-Based Strain Sensors: Achieving High Sensitivity and Wide Detection for Human Motion Detection and Wireless Transmission. ACS Sens. 2024 Apr 26;9(4):2156-2165. doi: 10.1021/acssensors.4c00274. Epub 2024 Apr 17. PMID 38629405
- [Background] Lin S, Pan X, Meng D, Zhang T. Electric conversion treatment of cobalt-containing wastewater. Water Sci Technol. 2021 Apr;83(8):1973-1986. doi: 10.2166/wst.2021.101. PMID 33905366
- [Background] Kawada T. Psychosocial factors and mortality in patients with heart failure. Eur J Heart Fail. 2018 Aug;20(8):1243. doi: 10.1002/ejhf.1208. Epub 2018 Apr 24. No abstract available. PMID 29693755
- [Background] Murphy HR, Howgate C, O'Keefe J, Myers J, Morgan M, Coleman MA, Jolly M, Valabhji J, Scott EM, Knighton P, Young B, Lewis-Barned N; National Pregnancy in Diabetes (NPID) advisory group. Characteristics and outcomes of pregnant women with type 1 or type 2 diabetes: a 5-year national population-based cohort study. Lancet Diabetes Endocrinol. 2021 Mar;9(3):153-164. doi: 10.1016/S2213-8587(20)30406-X. Epub 2021 Jan 28. PMID 33516295
- [Background] Simmons D, Immanuel J, Hague WM, Teede H, Nolan CJ, Peek MJ, Flack JR, McLean M, Wong V, Hibbert E, Kautzky-Willer A, Harreiter J, Backman H, Gianatti E, Sweeting A, Mohan V, Enticott J, Cheung NW; TOBOGM Research Group. Treatment of Gestational Diabetes Mellitus Diagnosed Early in Pregnancy. N Engl J Med. 2023 Jun 8;388(23):2132-2144. doi: 10.1056/NEJMoa2214956. Epub 2023 May 5. PMID 37144983